CLINICAL TRIAL: NCT00006089
Title: A Phase II Evaluation of Trastuzumab (MoAb HER2) in Patients With Advanced, Recurrent or Persistent Endometrial Carcinoma With or Without Prior Chemotherapy
Brief Title: Trastuzumab in Treating Patients With Stage III, Stage IV, or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02356; NCI-2012-02356 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068091; GOG-0181B; GOG-0181-B (Other: Gynecologic Oncology Group); GOG-0181B (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Endometrial Adenocarcinoma; ERBB2 Gene Amplification; Recurrent Uterine Corpus Carcinoma; Stage III Uterine Corpus Cancer AJCC v7; Stage IV Uterine Corpus Cancer AJCC v7
MeSH Terms: interventions — Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

ARMS (1):
- Treatment (trastuzumab) (Experimental): Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Trastuzumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab-dkst; Trastuzumab-DTTB; Trastuzumab-pkrb; Trastuzumab-QYYP; Trazimera

SUMMARY:
Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Phase II trial to study the effectiveness of trastuzumab in treating patients who have stage III, stage IV, or recurrent endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OOBJECTIVES:

I. Determine the antitumor activity of trastuzumab (Herceptin), in terms of response, in patients with advanced, recurrent, or persistent endometrial adenocarcinoma that demonstrates HER2/neu gene amplification by fluorescent in situ hybridization.

II. Determine the toxicity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the progression-free and overall survival of patients treated with this regimen.

II. Determine the effects of prognostic factors (i.e., initial performance status and histological grade) in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 25-42 patients will be accrued for this study within 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial adenocarcinoma

  * Advanced, recurrent, or persistent disease
  * Refractory to curative therapy
* HER2/neu gene amplification by fluorescent in situ hybridization
* Measurable disease

  * Previously irradiated field as sole site of measurable disease allowed if evidence of progression since completion of radiotherapy
* Performance status - GOG 0-2
* Absolute neutrophil count ? 1,500/mm^3
* Platelet count ? 100,000/mm^3
* Bilirubin ? 1.5 times upper limit of normal (ULN)
* Creatinine ? 1.5 times ULN
* LVEF ? 45% by echocardiogram or MUGA
* History of coronary artery disease and/or congestive heart failure allowed if medical management of condition has been stable within the past 6 months
* No active or unstable cardiac disease
* No active angina
* No myocardial infarction within the past 6 months
* No requirement for supplemental oxygen at rest or with ambulation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No uncontrolled infection
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No other unstable medical condition that would preclude study participation
* At least 3 weeks since prior biologic and immunologic agents directed at the malignant tumor
* No prior anti-HER2 monoclonal antibody preparation
* No other concurrent immunotherapy
* Recovered from prior chemotherapy
* Multiple prior chemotherapy regimens allowed
* No more than 320 mg/m^2 total dose of prior doxorubicin allowed (including doxorubicin HCl liposome or other liposomally encapsulated doxorubicin preparations)
* No concurrent chemotherapy
* At least 1 week since prior hormonal therapy directed at the malignant tumor
* No concurrent hormonal therapy

  * Continuation of hormone replacement therapy allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for the malignant tumor and recovered
* No concurrent radiotherapy
* Recovered from prior recent surgery
* At least 3 weeks since any prior therapy directed at the malignant tumor
* No prior cancer treatment that would contraindicate study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-09-18 (Actual); Primary Completion 2007-09-04 (Actual); Study Completion 2010-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency and duration of objective response | Up to 5 years
Frequency and severity of observed adverse effects assessed using Common Terminology Criteria (CTC) version 2.0 | Up to 5 years

SECONDARY OUTCOMES:
Duration of progression-free survival | From study entry until disease progression, death or date or last contact, assessed up to 5 years
  Will be evaluated with non-parametric statistics (such as the log-rank test) through comparisons with the historical controls.
Duration of overall survival | From study entry to death or date or last contact, assessed up to 5 years
  Will be evaluated with non-parametric statistics (such as the log-rank test) through comparisons with the historical controls.
Prognostic factors (i.e., initial performance status and histological grade) | Not Provided
  Comparisons will be made through a Cox model, which allows for adjustments with the prognostic variables.

CONTACTS AND LOCATIONS:
Overall Officials: Gini F Fleming, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States